CLINICAL TRIAL: NCT06942247
Title: A Clinical Study to Evaluate the Safety and Efficacy of Biologic Hollow Bone Screws
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Follow-up data for the last participant cannot be fully collected within the next year and cannot be entered on the website in time; therefore, we request approval to update the trial status to "Suspended."
Sponsor: FengYafei (Other)
Responsible Party: Sponsor-Investigator, FengYafei, Associate professor, Xijing Hospital
Organization: Xijing Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: QX20221007-X-1
Record Dates: First submitted 2024-04-28; First posted 2025-04-24 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Fracture Fixation, Internal
Keywords: Silk fibroin bone screws; Fracture fixation; Knee and ankle joints; Safety and efficacy evaluation; Prognosis

STUDY DESIGN:
Intervention Model Description: The experimental group was treated with biologic hollow bone screws (Jiangxi Sike Biotechnology, China); the control group was treated with Freedom Screws (Inion Oy, Finland).
Who Masked: Participant
Masking Description: The researchers can visually distinguish the experiment products and the control products, so the researchers cannot be blinded and the participants were blinded.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inion Freedom Screws (Active Comparator): Patients were treated with screws developed by Inion Oy, Finland for the fixation of fractures in the knee and ankle joints.
  Interventions: Device: Active Comparator: Fracture Fixation (Inion Freedom Screws)
- Biologic Hollow Bone Screws (Experimental): Patients were treated with screws developed by Jiangxi Sike Biotechnology, China for the fixation of fractures in the knee and ankle joints.
  Interventions: Device: Experimental: Fracture Fixation (Biological Hollow Bone Screws)

INTERVENTIONS:
Device: Active Comparator: Fracture Fixation (Inion Freedom Screws) — Device: Absorbable screw for internal fixation of fracture. Patients were divided into the Inion Freedom Screws group and the Biological Hollow Bone Screws group according to the type of the screws they used.
  Arms: Inion Freedom Screws
Device: Experimental: Fracture Fixation (Biological Hollow Bone Screws) — Device: Absorbable screw for internal fixation of fracture. Patients were divided into the Inion Freedom Screws group and the Biological Hollow Bone Screws group according to the type of the screws they used.
  Arms: Biologic Hollow Bone Screws

SUMMARY:
Traditional fracture fixation devices can cause corrosion, allergies, and stress shielding effects. They often require removal after healing, risking secondary damage. Recently, biodegradable materials have gained attention for their effective clinical use in fracture fixation. Absorbable bone nails, for example, eliminate the need for a second surgery, reducing pain and costs while avoiding infection and tissue re-injury. They do not corrode and are invisible on X-rays, allowing for thorough patient examination and better fracture healing assessment.

DETAILED DESCRIPTION:
Traditional fracture internal fixation devices implanted in the human body for a long time will cause corrosion, allergy and adverse effects due to stress shielding effect, etc. Due to the non-absorbability of its own materials, it needs to be removed again after fracture healing, which is easy to cause secondary damage to patients. However, in recent years, biodegradable materials have attracted the attention of scholars. The fracture fixation made of biodegradable biomaterials has achieved better internal fixation effect in clinic. For example, the implantation of absorbable bone nails can enable patients to avoid a second surgery, reduce the pain and economic burden of patients, while avoiding the problems of infection and tissue re-injury caused by the second surgery. In addition, absorbable bone nails have no metal corrosion effect and are not visible under the X-ray line, which is conducive to comprehensive examination of the patient and further understanding of the fracture healing. Common biodegradable materials are polymer materials (such as polylactic acid), ceramic materials (such as calcium phosphate) and metal materials. Among them, the strength of polymer materials is lower, and the toughness of ceramic materials is poorer, while the bone nails made of natural silk protein are biocompatible, non-toxic, no irritant, no side-effective, no antigenic and no carcinogenic to tissues. It can be completely degraded into amino acids and peptides in the body, participate in human metabolism, and eventually be excreted from the body. Silk was first used as a surgical suture, which can be gradually absorbed and degraded by the body after wound healing, which protected patients from the pain of removing stitches. Animal experiments have shown that the use of silk protein gel and commonly used ethyl lactate to repair rabbit thigh bone injuries, with the number, thickness and gap of bone trabeculae as evaluation indexes, the result showed that the use of silk protein gel was more conducive to the repair of rabbit thigh bone injury, and was also closer to the regeneration of human bone. In addition, the silk was able to maintain 50% tension two months after implantation in the animals.

Therefore, the purpose of this clinical trial study was to evaluate the safety and effectiveness of biologic hollow bone screws for the fixation of fractures in the knee joint and ankle joint. Researchers can use the above results to provide better treatment for patients.

ELIGIBILITY:
Inclusion criteria

1. Aged 18-75 years old (inclusive), both sexes;
2. Patients with knee and ankle fractures requiring internal fixation confirmed by imaging examination;
3. Voluntary participation in the clinical trial and signing of the informed consent.

Exclusion criteria

1. The following conditions exist at the fracture site: infection, osteofascial compartment syndrome, osteitis, pathological fracture, open fracture, severe tissue or vascular and nerve injury, or insufficient bone mass of the affected limb affecting screw implantation, etc.
2. Abnormal liver and kidney function with clinical significance (ALT, AST 2 times the upper limit of normal value and Cr 2 times the upper limit of normal value);
3. Abnormal coagulation function with clinical significance (APTT > 2 times the upper limit of normal value);
4. Patients with difficult-to-control diabetes (any blood glucose > 11.1mmol/L or glycosylated hemoglobin > 9%);
5. Past allergies to silk protein materials;
6. Mental illness;
7. Patients who cannot guarantee to quit smoking during the fracture healing period;
8. Pregnant or lactating women or women of childbearing age who plan to get pregnant within 6 months;
9. Those who have participated in other pre-clinical trials within 1 month before the trial;
10. Those who are considered inappropriate to participate in the clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Cinical Fracture Healing Rate | 24 weeks after surgery+4 weeks
  1. No local tenderness or longitudinal percussion pain, no local abnormal activity;
  2. X-rays show a continuous bone scab or trabeculae crossing the fracture line at the fracture site and the fracture line has been blurred. If both of these are met, the fracture is considered healed, and vice versa.
  3. Healing rate = (Healing cases / Total cases) ×100%

SECONDARY OUTCOMES:
Cinical Fracture Healing Rate | 12 weeks after surgery±1 week
  1. No local tenderness or longitudinal percussion pain, no local abnormal activity;
  2. X-rays show a continuous bone scab or trabeculae crossing the fracture line at the fracture site and the fracture line has been blurred. If both of these are met, the fracture is considered healed, and vice versa.
  3. Healing rate = (Healing cases / Total cases) ×100%
Cinical Fracture Healing Rate | 48 weeks after surgery± 4 weeks
  1. No local tenderness or longitudinal percussion pain, no local abnormal activity;
  2. X-rays show a continuous bone scab or trabeculae crossing the fracture line at the fracture site and the fracture line has been blurred. If both of these are met, the fracture is considered healed, and vice versa.
  3. Healing rate = (Healing cases / Total cases) ×100%
Cinical Fracture Healing Rate | 72 weeks after surgery± 4 weeks
  1. No local tenderness or longitudinal percussion pain, no local abnormal activity;
  2. X-rays show a continuous bone scab or trabeculae crossing the fracture line at the fracture site and the fracture line has been blurred. If both of these are met, the fracture is considered healed, and vice versa.
  3. Healing rate = (Healing cases / Total cases) ×100%
Visual Analogue Scale (VAS) | During the screening period
  In the Visual Analogue Scale (VAS), the minimum value is 0 and the maximum value is 10. The higher the score, the more severe the pain and the worse the outcome.
  A score of 0 means painless; A score of 1-3 means mild pain, tolerable; A score of 4-6 indicates moderate pain that affects sleep and is tolerable; A score of 7-10 indicates severe pain, unbearable pain, affecting appetite, and affecting sleep.
Visual Analogue Scale (VAS) | Within 1 week after surgery (≤7 days)
  In the Visual Analogue Scale (VAS), the minimum value is 0 and the maximum value is 10. The higher the score, the more severe the pain and the worse the outcome.
  A score of 0 means painless; A score of 1-3 means mild pain, tolerable; A score of 4-6 indicates moderate pain that affects sleep and is tolerable; A score of 7-10 indicates severe pain, unbearable pain, affecting appetite, and affecting sleep.
Visual Analogue Scale (VAS) | 6 weeks after surgery±1 week
  In the Visual Analogue Scale (VAS), the minimum value is 0 and the maximum value is 10. The higher the score, the more severe the pain and the worse the outcome.
  A score of 0 means painless; A score of 1-3 means mild pain, tolerable; A score of 4-6 indicates moderate pain that affects sleep and is tolerable; A score of 7-10 indicates severe pain, unbearable pain, affecting appetite, and affecting sleep.
Visual Analogue Scale (VAS) | 12 weeks after surgery±1 week
  In the Visual Analogue Scale (VAS), the minimum value is 0 and the maximum value is 10. The higher the score, the more severe the pain and the worse the outcome.
  A score of 0 means painless; A score of 1-3 means mild pain, tolerable; A score of 4-6 indicates moderate pain that affects sleep and is tolerable; A score of 7-10 indicates severe pain, unbearable pain, affecting appetite, and affecting sleep.
Visual Analogue Scale (VAS) | 24 weeks after surgery±4 weeks
  In the Visual Analogue Scale (VAS), the minimum value is 0 and the maximum value is 10. A higher score indicates a more severe level of pain.
  A score of 0 means painless; A score of 1-3 means mild pain, tolerable; A score of 4-6 indicates moderate pain that affects sleep and is tolerable; A score of 7-10 indicates severe pain, unbearable pain, affecting appetite, and affecting sleep.
Visual Analogue Scale (VAS) | 48 weeks after surgery±4 weeks
  In the Visual Analogue Scale (VAS), the minimum value is 0 and the maximum value is 10. The higher the score, the more severe the pain and the worse the outcome.
  A score of 0 means painless; A score of 1-3 means mild pain, tolerable; A score of 4-6 indicates moderate pain that affects sleep and is tolerable; A score of 7-10 indicates severe pain, unbearable pain, affecting appetite, and affecting sleep.
Visual Analogue Scale (VAS) | 72 weeks after surgery± 4 weeks
  In the Visual Analogue Scale (VAS), the minimum value is 0 and the maximum value is 10. The higher the score, the more severe the pain and the worse the outcome.
  A score of 0 means painless; A score of 1-3 means mild pain, tolerable; A score of 4-6 indicates moderate pain that affects sleep and is tolerable; A score of 7-10 indicates severe pain, unbearable pain, affecting appetite, and affecting sleep.
The American Knee Society (AKS) Clinical Rating System | 6 weeks after surgery±1 week
  AKS score is divided into two parts: knee score and functional score. The knee score includes pain, range of motion and stability, and the functional score includes the ability to walk and go up and down stairs.
  The knee score is an assessment of knee pain, stability, and range of motion. And the functional score is an assessment of walking ability and the ability to walk up and down stairs.
  The total score of AKS is 200 points, of which knee score and functional score are 100 points each. The higher the score, the better the status. If the score is negative, it is calculated as 0.
The American Knee Society (AKS) Clinical Rating System | 12 weeks after surgery±1 week
  AKS score is divided into two parts: knee score and functional score. The knee score includes pain, range of motion and stability, and the functional score includes the ability to walk and go up and down stairs.
  The knee score is an assessment of knee pain, stability, and range of motion. And the functional score is an assessment of walking ability and the ability to walk up and down stairs.
  The total score of AKS is 200 points, of which knee score and functional score are 100 points each. The higher the score, the better the status. If the score is negative, it is calculated as 0.
The American Knee Society (AKS) Clinical Rating System | 24 weeks after surgery±4 weeks
  AKS score is divided into two parts: knee score and functional score. The knee score includes pain, range of motion and stability, and the functional score includes the ability to walk and go up and down stairs.
  The knee score is an assessment of knee pain, stability, and range of motion. And the functional score is an assessment of walking ability and the ability to walk up and down stairs.
  The total score of AKS is 200 points, of which knee score and functional score are 100 points each. The higher the score, the better the status. If the score is negative, it is calculated as 0.
The American Knee Society (AKS) Clinical Rating System | 48 weeks after surgery±4 weeks
  AKS score is divided into two parts: knee score and functional score. The knee score includes pain, range of motion and stability, and the functional score includes the ability to walk and go up and down stairs.
  The knee score is an assessment of knee pain, stability, and range of motion. And the functional score is an assessment of walking ability and the ability to walk up and down stairs.
  The total score of AKS is 200 points, of which knee score and functional score are 100 points each. The higher the score, the better the status. If the score is negative, it is calculated as 0.
The American Knee Society (AKS) Clinical Rating System | 72 weeks after surgery± 4 weeks
  AKS score is divided into two parts: knee score and functional score. The knee score includes pain, range of motion and stability, and the functional score includes the ability to walk and go up and down stairs.
  The knee score is an assessment of knee pain, stability, and range of motion. And the functional score is an assessment of walking ability and the ability to walk up and down stairs.
  The total score of AKS is 200 points, of which knee score and functional score are 100 points each. The higher the score, the better the status. If the score is negative, it is calculated as 0.
Mazur Ankle Joint Functional Evaluation | 6 weeks after surgery±1 week
  On the Mazur ankle joint functional evaluation, the highest score is 100, and a higher score indicates better ankle function.
  Excellent: >92 points, ankle joint without swelling pain, normal gait, free movement.
  Good: 87-92 points, ankle joint slight swelling pain, normal gait, range of motion up to 3/4 of normal.
  General: 65-86 points, pain during activity, only 1/2 of normal motion, normal gait, need to take non-steroidal anti-inflammatory drugs.
  Poor: <65 points, walking or resting pain, only 1/2 of normal range of motion, claudication, swollen ankle.
Mazur Ankle Joint Functional Evaluation | 12 weeks after surgery±1 week
  On the Mazur ankle joint functional evaluation, the highest score is 100, and a higher score indicates better ankle function.
  Excellent: >92 points, ankle joint without swelling pain, normal gait, free movement.
  Good: 87-92 points, ankle joint slight swelling pain, normal gait, range of motion up to 3/4 of normal.
  General: 65-86 points, pain during activity, only 1/2 of normal motion, normal gait, need to take non-steroidal anti-inflammatory drugs.
  Poor: <65 points, walking or resting pain, only 1/2 of normal range of motion, claudication, swollen ankle.
Mazur Ankle Joint Functional Evaluation | 24 weeks after surgery±4 weeks
  On the Mazur ankle joint functional evaluation, the highest score is 100, and a higher score indicates better ankle function.
  Excellent: >92 points, ankle joint without swelling pain, normal gait, free movement.
  Good: 87-92 points, ankle joint slight swelling pain, normal gait, range of motion up to 3/4 of normal.
  General: 65-86 points, pain during activity, only 1/2 of normal motion, normal gait, need to take non-steroidal anti-inflammatory drugs.
  Poor: <65 points, walking or resting pain, only 1/2 of normal range of motion, claudication, swollen ankle.
Mazur Ankle Joint Functional Evaluation | 48 weeks after surgery±4 weeks
  On the Mazur ankle joint functional evaluation, the highest score is 100, and a higher score indicates better ankle function.
  Excellent: >92 points, ankle joint without swelling pain, normal gait, free movement.
  Good: 87-92 points, ankle joint slight swelling pain, normal gait, range of motion up to 3/4 of normal.
  General: 65-86 points, pain during activity, only 1/2 of normal motion, normal gait, need to take non-steroidal anti-inflammatory drugs.
  Poor: <65 points, walking or resting pain, only 1/2 of normal range of motion, claudication, swollen ankle.
Mazur Ankle Joint Functional Evaluation | 72 weeks after surgery± 4 weeks
  On the Mazur ankle joint functional evaluation, the highest score is 100, and a higher score indicates better ankle function.
  Excellent: >92 points, ankle joint without swelling pain, normal gait, free movement.
  Good: 87-92 points, ankle joint slight swelling pain, normal gait, range of motion up to 3/4 of normal.
  General: 65-86 points, pain during activity, only 1/2 of normal motion, normal gait, need to take non-steroidal anti-inflammatory drugs.
  Poor: <65 points, walking or resting pain, only 1/2 of normal range of motion, claudication, swollen ankle.

OTHER OUTCOMES:
Demographic Data | Before surgery
  It mainly includes the age, gender, place of birth and education level of the patient
History of Disease and Treatment | Before surgery
  Medical history within 3 months before signing the informed consent, medication history, surgery history, smoking history, drinking history and allergy history within 1 month before signing the informed consent were asked.
Bone Mineral Density (BMD) Examination | Before surgery
  Bone Mineral Density (BMD) Examination
Blood Glucose Testing | Before surgery
  Blood Glucose Testing
C-Reactive Protein | Before surgery
  C-Reactive Protein
Examination of Infectious Diseases | Before surgery
  Hepatitis B Surface Antigen (HBsAg)
Examination of Infectious Diseases | Before surgery
  Hepatitis B Surface Antibody (HBsAb)
Examination of Infectious Diseases | Before surgery
  Hepatitis B e-Antigen (HBeAg)
Examination of Infectious Diseases | Before surgery
  Hepatitis B e-Antibody (HBeAb)
Examination of Infectious Diseases | Before surgery
  Hepatitis B Core Antibody (HBcAb)
Examination of Infectious Diseases | Before surgery
  Hepatitis Virus C-RNA / Hepatitis Virus C-Antibody (HCV-rna/HCV-Ab)
Examination of Infectious Diseases | Before surgery
  Treponema Pallidum Particle Agglutination Assay (TPPA)
Examination of Infectious Diseases | Before surgery
  Human Immunodeficiency Virus Antibody (HIV-Ab)
Record Surgical Information | During Surgery
  Operation time
Record Surgical Information | During Surgery
  Intraoperative blood loss
Record Surgical Information | During Surgery
  Device usage
Vital Signs-Body Temperature | Before surgery
  Body Temperature
Vital Signs-Respiration | Before surgery
  Respiration
Vital Signs-Heart Rate | Before surgery
  Heart Rate
Vital Signs-Blood Pressure | Before surgery
  Blood Pressure
Vital Signs-Body Temperature | During Surgery
  Body Temperature
Vital Signs-Respiration | During Surgery
  Respiration
Vital Signs-Heart Rate | During Surgery
  Heart Rate
Vital Signs-Blood Pressure | During Surgery
  Blood Pressure
Vital Signs-Body Temperature | Within 1 week after surgery (≤7 days)
  Body Temperature
Vital Signs-Respiration | Within 1 week after surgery (≤7 days)
  Respiration
Vital Signs-Heart Rate | Within 1 week after surgery (≤7 days)
  Heart Rate
Vital Signs-Blood Pressure | Within 1 week after surgery (≤7 days)
  Blood Pressure
Vital Signs-Body Temperature | 6 weeks after surgery±1 week
  Body Temperature
Vital Signs-Respiration | 6 weeks after surgery±1 week
  Respiration
Vital Signs-Heart Rate | 6 weeks after surgery±1 week
  Heart Rate
Vital Signs-Blood Pressure | 6 weeks after surgery±1 week
  Blood Pressure
Vital Signs-Body Temperature | 12 weeks after surgery±1 week
  Body Temperature
Vital Signs-Respiration | 12 weeks after surgery±1 week
  Respiration
Vital Signs-Heart Rate | 12 weeks after surgery±1 week
  Heart Rate
Vital Signs-Blood Pressure | 12 weeks after surgery±1 week
  Blood Pressure
Vital Signs-Body Temperature | 24 weeks after surgery±4 weeks
  Body Temperature
Vital Signs-Respiration | 24 weeks after surgery±4 weeks
  Respiration
Vital Signs-Heart Rate | 24 weeks after surgery±4 weeks
  Heart Rate
Vital Signs-Blood Pressure | 24 weeks after surgery±4 weeks
  Blood Pressure
Vital Signs-Body Temperature | 48 weeks after surgery±4 weeks
  Body Temperature
Vital Signs-Respiration | 48 weeks after surgery±4 weeks
  Respiration
Vital Signs-Heart Rate | 48 weeks after surgery±4 weeks
  Heart Rate
Vital Signs-Blood Pressure | 48 weeks after surgery±4 weeks
  Blood Pressure
Vital Signs-Body Temperature | 72 weeks after surgery± 4 weeks
  Body Temperature
Vital Signs-Respiration | 72 weeks after surgery± 4 weeks
  Respiration
Vital Signs-Heart Rate | 72 weeks after surgery± 4 weeks
  Heart Rate
Vital Signs-Blood Pressure | 72 weeks after surgery± 4 weeks
  Blood Pressure
Laboratory Examinations-X-Ray Examination | During the screening period
  X-Ray Examination
Laboratory Examinations-X-Ray Examination | Within 1 week after surgery (≤7 days)
  X-Ray Examination
Laboratory Examinations-X-Ray Examination | 6 weeks after surgery±1 week
  X-Ray Examination
Laboratory Examinations-X-Ray Examination | 12 weeks after surgery±1 week
  X-Ray Examination
Laboratory Examinations-X-Ray Examination | 24 weeks after surgery±4 weeks
  X-Ray Examination
Laboratory Examinations-X-Ray Examination | 48 weeks after surgery±4 weeks
  X-Ray Examination
Laboratory Examinations-X-Ray Examination | 72 weeks after surgery±4 weeks
  X-Ray Examination
Laboratory Examinations-Coagulation Function | During the screening period
  Prothrombin Time (PT)
Laboratory Examinations-Coagulation Function | During the screening period
  Activated Partial Thromboplastin Time (APTT)
Laboratory Examinations-Coagulation Function | During the screening period
  Fibrinogen (FIB)
Laboratory Examinations-Coagulation Function | During the screening period
  Thrombin Time (TT)
Laboratory Examinations-Coagulation Function | Within 1 week after surgery (≤7 days)
  Prothrombin Time (PT)
Laboratory Examinations-Coagulation Function | Within 1 week after surgery (≤7 days)
  Activated Partial Thromboplastin Time (APTT)
Laboratory Examinations-Coagulation Function | Within 1 week after surgery (≤7 days)
  Fibrinogen (FIB)
Laboratory Examinations-Coagulation Function | Within 1 week after surgery (≤7 days)
  Thrombin Time (TT)
Laboratory Examinations-Coagulation Function | 24 weeks after surgery±4 weeks
  Prothrombin Time (PT)
Laboratory Examinations-Coagulation Function | 24 weeks after surgery±4 weeks
  Activated Partial Thromboplastin Time (APTT)
Laboratory Examinations-Coagulation Function | 24 weeks after surgery±4 weeks
  Fibrinogen (FIB)
Laboratory Examinations-Coagulation Function | 24 weeks after surgery±4 weeks
  Thrombin Time (TT)
Laboratory Examinations-Coagulation Function | 48 weeks after surgery±4 weeks
  Prothrombin Time (PT)
Laboratory Examinations-Coagulation Function | 48 weeks after surgery±4 weeks
  Activated Partial Thromboplastin Time (APTT)
Laboratory Examinations-Coagulation Function | 48 weeks after surgery±4 weeks
  Fibrinogen (FIB)
Laboratory Examinations-Coagulation Function | 48 weeks after surgery±4 weeks
  Thrombin Time (TT)
Laboratory Examinations-Coagulation Function | 72 weeks after surgery±4 weeks
  Prothrombin Time (PT)
Laboratory Examinations-Coagulation Function | 72 weeks after surgery±4 weeks
  Activated Partial Thromboplastin Time (APTT)
Laboratory Examinations-Coagulation Function | 72 weeks after surgery±4 weeks
  Fibrinogen (FIB)
Laboratory Examinations-Coagulation Function | 72 weeks after surgery±4 weeks
  Thrombin Time (TT)
Laboratory Examinations-Routine Blood Test | During the screening period
  Hemoglobin (Hb)
Laboratory Examinations-Routine Blood Test | During the screening period
  Red Blood Cell Count (RBC)
Laboratory Examinations-Routine Blood Test | During the screening period
  White Blood Cell Count (WBC)
Laboratory Examinations-Routine Blood Test | During the screening period
  Platelet Count (PLT)
Laboratory Examinations-Routine Blood Test | During the screening period
  Hematocrit (HCT)
Laboratory Examinations-Routine Blood Test | Within 1 week after surgery (≤7 days)
  Hemoglobin (Hb)
Laboratory Examinations-Routine Blood Test | Within 1 week after surgery (≤7 days)
  Red Blood Cell Count (RBC)
Laboratory Examinations-Routine Blood Test | Within 1 week after surgery (≤7 days)
  White Blood Cell Count (WBC)
Laboratory Examinations-Routine Blood Test | Within 1 week after surgery (≤7 days)
  Platelet Count (PLT)
Laboratory Examinations-Routine Blood Test | Within 1 week after surgery (≤7 days)
  Hematocrit (HCT)
Laboratory Examinations-Routine Blood Test | 24 weeks after surgery± 4 weeks
  Hemoglobin (Hb)
Laboratory Examinations-Routine Blood Test | 24 weeks after surgery± 4 weeks
  Red Blood Cell Count (RBC)
Laboratory Examinations-Routine Blood Test | 24 weeks after surgery± 4 weeks
  White Blood Cell Count (WBC)
Laboratory Examinations-Routine Blood Test | 24 weeks after surgery± 4 weeks
  Platelet Count (PLT)
Laboratory Examinations-Routine Blood Test | 24 weeks after surgery± 4 weeks
  Hematocrit (HCT)
Laboratory Examinations-Routine Blood Test | 48 weeks after surgery± 4 weeks
  Hemoglobin (Hb)
Laboratory Examinations-Routine Blood Test | 48 weeks after surgery± 4 weeks
  Red Blood Cell Count (RBC)
Laboratory Examinations-Routine Blood Test | 48 weeks after surgery± 4 weeks
  White Blood Cell Count (WBC)
Laboratory Examinations-Routine Blood Test | 48 weeks after surgery± 4 weeks
  Platelet Count (PLT)
Laboratory Examinations-Routine Blood Test | 48 weeks after surgery± 4 weeks
  Hematocrit (HCT)
Laboratory Examinations-Routine Blood Test | 72 weeks after surgery± 4 weeks
  Hemoglobin (Hb)
Laboratory Examinations-Routine Blood Test | 72 weeks after surgery± 4 weeks
  Red Blood Cell Count (RBC)
Laboratory Examinations-Routine Blood Test | 72 weeks after surgery± 4 weeks
  White Blood Cell Count (WBC)
Laboratory Examinations-Routine Blood Test | 72 weeks after surgery± 4 weeks
  Platelet Count (PLT)
Laboratory Examinations-Routine Blood Test | 72 weeks after surgery± 4 weeks
  Hematocrit (HCT)
Laboratory Examinations-Routine Urine Test | During the screening period
  Urine Protein (PRO)
Laboratory Examinations-Routine Urine Test | During the screening period
  Urine Red Blood Cells (RBC)
Laboratory Examinations-Routine Urine Test | During the screening period
  Urine Glucose (GLU)
Laboratory Examinations-Routine Urine Test | Within 1 week after surgery (≤7 days)
  Urine Protein (PRO)
Laboratory Examinations-Routine Urine Test | Within 1 week after surgery (≤7 days)
  Urine Red Blood Cells (RBC)
Laboratory Examinations-Routine Urine Test | Within 1 week after surgery (≤7 days)
  Urine Glucose (GLU)
Laboratory Examinations-Routine Urine Test | 24 weeks after surgery± 4 weeks
  Urine Protein (PRO)
Laboratory Examinations-Routine Urine Test | 24 weeks after surgery± 4 weeks
  Urine Red Blood Cells (RBC)
Laboratory Examinations-Routine Urine Test | 24 weeks after surgery± 4 weeks
  Urine Glucose (GLU)
Laboratory Examinations-Routine Urine Test | 48 weeks after surgery± 4 weeks
  Urine Protein (PRO)
Laboratory Examinations-Routine Urine Test | 48 weeks after surgery± 4 weeks
  Urine Red Blood Cells (RBC)
Laboratory Examinations-Routine Urine Test | 48 weeks after surgery± 4 weeks
  Urine Glucose (GLU)
Laboratory Examinations-Routine Urine Test | 72 weeks after surgery± 4 weeks
  Urine Protein (PRO)
Laboratory Examinations-Routine Urine Test | 72 weeks after surgery± 4 weeks
  Urine Red Blood Cells (RBC)
Laboratory Examinations-Routine Urine Test | 72 weeks after surgery± 4 weeks
  Urine Glucose (GLU)
Laboratory Examinations-Blood Biochemical Examination | During the screening period
  Creatinine (Cr)
Laboratory Examinations-Blood Biochemical Examination | During the screening period
  Urea nitrogen (BUN)
Laboratory Examinations-Blood Biochemical Examination | During the screening period
  Urea (UREA)
Laboratory Examinations-Blood Biochemical Examination | During the screening period
  Alanine aminotransferase (ALT) / Aspartate aminotransferase (AST)
Laboratory Examinations-Blood Biochemical Examination | Within 1 week after surgery (≤7 days)
  Creatinine (Cr)
Laboratory Examinations-Blood Biochemical Examination | Within 1 week after surgery (≤7 days)
  Urea nitrogen (BUN)
Laboratory Examinations-Blood Biochemical Examination | Within 1 week after surgery (≤7 days)
  Urea (UREA)
Laboratory Examinations-Blood Biochemical Examination | Within 1 week after surgery (≤7 days)
  Alanine aminotransferase (ALT) / Aspartate aminotransferase (AST)
Laboratory Examinations-Blood Biochemical Examination | 24 weeks after surgery± 4 weeks
  Creatinine (Cr)
Laboratory Examinations-Blood Biochemical Examination | 24 weeks after surgery± 4 weeks
  Urea nitrogen (BUN)
Laboratory Examinations-Blood Biochemical Examination | 24 weeks after surgery± 4 weeks
  Urea (UREA)
Laboratory Examinations-Blood Biochemical Examination | 24 weeks after surgery± 4 weeks
  Alanine aminotransferase (ALT) / Aspartate aminotransferase (AST)
Laboratory Examinations-Blood Biochemical Examination | 48 weeks after surgery± 4 weeks
  Creatinine (Cr)
Laboratory Examinations-Blood Biochemical Examination | 48 weeks after surgery± 4 weeks
  Urea nitrogen (BUN)
Laboratory Examinations-Blood Biochemical Examination | 48 weeks after surgery± 4 weeks
  Urea (UREA)
Laboratory Examinations-Blood Biochemical Examination | 48 weeks after surgery± 4 weeks
  Alanine aminotransferase (ALT) / Aspartate aminotransferase (AST)
Laboratory Examinations-Blood Biochemical Examination | 72 weeks after surgery± 4 weeks
  Creatinine (Cr)
Laboratory Examinations-Blood Biochemical Examination | 72 weeks after surgery± 4 weeks
  Urea nitrogen (BUN)
Laboratory Examinations-Blood Biochemical Examination | 72 weeks after surgery± 4 weeks
  Urea (UREA)
Laboratory Examinations-Blood Biochemical Examination | 72 weeks after surgery± 4 weeks
  Alanine aminotransferase (ALT) / Aspartate aminotransferase (AST)
Defects of Device | During the screening period
  In the process of clinical trials, there are unreasonable risks of medical devices that may endanger human health and life safety under normal use, such as labeling errors, quality problems and malfunctions. In the course of this clinical trial, if the device fails due to the defect of the device, the investigator will carry out routine treatment according to clinical needs. Investigators should document all device discoveries that occur during the course of the clinical trial Defects.
Defects of Device | Before Surgery
  In the process of clinical trials, there are unreasonable risks of medical devices that may endanger human health and life safety under normal use, such as labeling errors, quality problems and malfunctions. In the course of this clinical trial, if the device fails due to the defect of the device, the investigator will carry out routine treatment according to clinical needs. Investigators should document all device discoveries that occur during the course of the clinical trial Defects.
Defects of Device | Within 1 week after surgery (≤7 days)
  In the process of clinical trials, there are unreasonable risks of medical devices that may endanger human health and life safety under normal use, such as labeling errors, quality problems and malfunctions. In the course of this clinical trial, if the device fails due to the defect of the device, the investigator will carry out routine treatment according to clinical needs. Investigators should document all device discoveries that occur during the course of the clinical trial Defects.
Defects of Device | 6 weeks after surgery±1 week
  In the process of clinical trials, there are unreasonable risks of medical devices that may endanger human health and life safety under normal use, such as labeling errors, quality problems and malfunctions. In the course of this clinical trial, if the device fails due to the defect of the device, the investigator will carry out routine treatment according to clinical needs. Investigators should document all device discoveries that occur during the course of the clinical trial Defects.
Defects of Device | 12 weeks after surgery±1 week
  In the process of clinical trials, there are unreasonable risks of medical devices that may endanger human health and life safety under normal use, such as labeling errors, quality problems and malfunctions. In the course of this clinical trial, if the device fails due to the defect of the device, the investigator will carry out routine treatment according to clinical needs. Investigators should document all device discoveries that occur during the course of the clinical trial Defects.
Defects of Device | 24 weeks after surgery±4 weeks
  In the process of clinical trials, there are unreasonable risks of medical devices that may endanger human health and life safety under normal use, such as labeling errors, quality problems and malfunctions. In the course of this clinical trial, if the device fails due to the defect of the device, the investigator will carry out routine treatment according to clinical needs. Investigators should document all device discoveries that occur during the course of the clinical trial Defects.
Defects of Device | 48 weeks after surgery±4 weeks
  In the process of clinical trials, there are unreasonable risks of medical devices that may endanger human health and life safety under normal use, such as labeling errors, quality problems and malfunctions. In the course of this clinical trial, if the device fails due to the defect of the device, the investigator will carry out routine treatment according to clinical needs. Investigators should document all device discoveries that occur during the course of the clinical trial Defects.
Defects of Device | 72 weeks after surgery± 4 weeks
  In the process of clinical trials, there are unreasonable risks of medical devices that may endanger human health and life safety under normal use, such as labeling errors, quality problems and malfunctions. In the course of this clinical trial, if the device fails due to the defect of the device, the investigator will carry out routine treatment according to clinical needs. Investigators should document all device discoveries that occur during the course of the clinical trial Defects.
Safety Parameters-Adverse Events | Before Surgery
  During screening or follow-up, subjects were not counted as serious adverse events for anticipated or scheduled procedures.
Safety Parameters-Adverse Events | Within 1 week after surgery (≤7 days)
  During screening or follow-up, subjects were not counted as serious adverse events for anticipated or scheduled procedures.
Safety Parameters-Adverse Events | 6 weeks after surgery±1 week
  During screening or follow-up, subjects were not counted as serious adverse events for anticipated or scheduled procedures.
Safety Parameters-Adverse Events | 12 weeks after surgery±1 week
  During screening or follow-up, subjects were not counted as serious adverse events for anticipated or scheduled procedures.
Safety Parameters-Adverse Events | 24 weeks after surgery±4 weeks
  During screening or follow-up, subjects were not counted as serious adverse events for anticipated or scheduled procedures.
Safety Parameters-Adverse Events | 48 weeks after surgery±4 weeks
  During screening or follow-up, subjects were not counted as serious adverse events for anticipated or scheduled procedures.
Safety Parameters-Adverse Events | 72 weeks after surgery± 4 weeks
  During screening or follow-up, subjects were not counted as serious adverse events for anticipated or scheduled procedures.
Drug Combination | During the screening period
  The relevant drugs other than glucose, normal saline and narcotic drugs used during the trial were recorded.
Drug Combination | Before Surgery
  The relevant drugs other than glucose, normal saline and narcotic drugs used during the trial were recorded.
Drug Combination | Within 1 week after surgery (≤7 days)
  The relevant drugs other than glucose, normal saline and narcotic drugs used during the trial were recorded.
Drug Combination | 6 weeks after surgery±1 week
  The relevant drugs other than glucose, normal saline and narcotic drugs used during the trial were recorded.
Drug Combination | 12 weeks after surgery±1 week
  The relevant drugs other than glucose, normal saline and narcotic drugs used during the trial were recorded.
Drug Combination | 24 weeks after surgery±4 weeks
  The relevant drugs other than glucose, normal saline and narcotic drugs used during the trial were recorded.
Drug Combination | 48 weeks after surgery±4 weeks
  The relevant drugs other than glucose, normal saline and narcotic drugs used during the trial were recorded.
Drug Combination | 72 weeks after surgery±4 weeks
  The relevant drugs other than glucose, normal saline and narcotic drugs used during the trial were recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Air Force Medical University (Xijing Hospital), Xi'an, Shaanxi, China

DOCUMENTS (2):
  • Study Protocol (2024-01-21): https://cdn.clinicaltrials.gov/large-docs/47/NCT06942247/Prot_000.pdf
  • Statistical Analysis Plan (2024-01-21): https://cdn.clinicaltrials.gov/large-docs/47/NCT06942247/SAP_001.pdf